CLINICAL TRIAL: NCT07047170
Title: Do Adults' Physical Activity Levels Effect Their Perceptions of Benefits/Barriers to Exercise and Their Perceptions of Physical Self
Brief Title: Impact of Physical Activity on Exercise Perceptions and Physical Self in Adults
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Collaborators: Uskudar University (Other)
Responsible Party: Principal Investigator, Elif Önder, Physical therapist, Istinye University
Other Study IDs: 2020/666
Record Dates: First submitted 2025-05-21; First posted 2025-07-02 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Health Behavior; Healthy Persons; Exercise; Exercise Adherence; Physical Activity in Adults; Physical Activity Maintenance; Self Concept
Keywords: health behavior; healthy persons; exercise; exercise adherence; benefit of exercise; barriers of exercise; self concept
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Minimal Active Group (MAG): Minimal Active Group
- Group 2: Inactive Group (IG): Inactive Group
- Group 3: Very Active Group (CAG): Very Active Group

SUMMARY:
The purpose of this observational study was to investigate whether the perceived benefits/barriers of exercise and physical self-perception of healthy adults with different physical activity levels differ. The main questions it aims to answer are:

1. Do healthy adults with different physical activity levels have different perceptions of exercise benefits/barriers?
2. Are there differences in physical self-perception of healthy adults with different physical activity levels? After being asked about their demographic information, healthy adults answered questions from the International Physical Activity Questionnaire, the Perception of Exercise Benefits/Barriers Questionnaire, and the Physical Self-perception Questionnaire.

DETAILED DESCRIPTION:
The sample size of the study was calculated as 384 with a power of 95% and a margin of error of 0.05. Individuals over the age of 18, who volunteer to participate in the study, accept the consent form, and can use a computer and/or mobile phone will participate in the study. The study will be conducted by filling out an online form using social media, e-mail, and other communication channels due to the social isolation process. Individuals will be asked questions such as age, gender, height, weight, marital status, whether they are employed, their profession, educational status, and exercise habits as stated in the socio-demographic information form.

The International Physical Activity Survey Short Form (IPAC) presented in the appendix will be used for the activities of individuals. Physical Activity level is determined in 3 categories; Category I: Inactive ones: <600 MET-min/wk Category II: Minimum Active: >600 - 3000 MET-min/wk Category III: HEPA active ones: <3000 MET-min/wk

Individuals' perceptions of exercise benefits/barriers will be assessed with the Exercise Benefit/Barrier Scale. The scale consists of a total of 43 items. The scale has 4 answers in the conditioned-choice Likert scale format, from 4 (strongly agree) to 1 (strongly disagree). The total score of the scale varies between 43-172. The scale has two subgroups, the Exercise Barrier Scale and the Exercise Benefit Scale. Each subgroup can be used independently. The score range of the benefit scale is between 29-116, and the score range of the barrier scale is between 14-56. The sum of all items in the scale gives the total score of the Exercise Benefit/Barrier scale. The higher the total scale score, the more the individual understands the benefits of exercise. The validity and reliability of this scale in Turkey was performed by Ortabağ, Ceylan, Akyüz and Bebiş.

The self-perception inventory will be used for individuals' self-perception. The inventory, which measures the person's 4 sub-dimensions (Athletic competence, physical condition, body attractiveness, strength) and general physical competence, consists of a total of 30 items, each sub-scale containing 6 items. The adaptation study of this inventory to Turkey was conducted by Aşçı and colleagues. For each item, the inventory presents the person with statements describing two different people and asks the person to determine the degree to which they resemble each of them. After first deciding which of the two different groups of people they resemble the most, the person grades this similarity using the expressions "Just right for me" or "Quite right for me". Scoring and calculation of the self-perception inventory; the items are scored between 1 and 4. "4" represents high competence, and "1" represents low competence. The inventory gives scores ranging from 6 to 24 in 5 different dimensions of physical perception.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18-65 ages

Exclusion Criteria:

* professional sports person,
* have a cognitive problems,
* having a recent surgical operation
* were in COVID-19 quarantine,
* have a health problem that could affect their physical activity level,
* BMI > 35 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adult persons
Sampling Method: Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The International Physical Activity Questionnaire-Short Form | 7 days
  The International Physical Activity Questionnaire-Short Form determined the participants' physical activity levels .
The Exercise Benefit/Barrier Scale | 7 days
  The Exercise Benefit/Barrier Scale measured participants' perceptions of benefits and barriers to exercise
The Physical Self-Perception Profile (PSPP) | 7 days
  The Physical Self-Perception Profile (PSPP) was used to evaluate the participants' physical self-perception.

CONTACTS AND LOCATIONS:
Overall Officials: elif önder, Study Director — Istinye University
Locations (2):
- Turkey (Türkiye) (2):
  - Ondokuz Mayıs Üniversitesi, SUVAM Havza Fizik Tedavi ve Rehabilitasyon Merkezin, Samsun, Havza
  - Social Media, Samsun

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Prijatelj, K., Selak Bagarić, E., & Buljan Flander, G. (2022). Examination of Some Predictors of One's Physical Appearance, Life-Satisfaction and Self-Esteem in the Wider Context of Engaging in Fitness Programs. Socijalne teme: Časopis za pitanja socijalnog rada i srodnih znanosti, 1(9), 25-46.
- [Result] Pulido JJ, Tapia-Serrano MA, Diaz-Garcia J, Ponce-Bordon JC, Lopez-Gajardo MA. The Relationship between Students' Physical Self-Concept and Their Physical Activity Levels and Sedentary Behavior: The Role of Students' Motivation. Int J Environ Res Public Health. 2021 Jul 22;18(15):7775. doi: 10.3390/ijerph18157775. PMID 34360069
- [Result] Schilling R, Schmidt SCE, Fiedler J, Woll A. Associations between physical activity, physical fitness, and body composition in adults living in Germany: A cross-sectional study. PLoS One. 2023 Oct 26;18(10):e0293555. doi: 10.1371/journal.pone.0293555. eCollection 2023. PMID 37883524

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT07047170/Prot_SAP_000.pdf